CLINICAL TRIAL: NCT01667393
Title: Popliteal Artery Trial of Patients Undergoing Treatment With Balloon Angioplasty vs. the Adaptive SUPERA VERITAS Peripheral Stent System
Brief Title: Popliteal Artery of Treatment With Balloon Angioplasty vs. SUPERA VERITAS Peripheral Stent System
Acronym: PARADIGM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDEV POP-01-US/OUS
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDEV SUPERA Stent (Experimental): Following PTA of the target lesion, the SUPERA stent will be delivered to the treated segment.
  Interventions: Device: IDEV SUPERA Stent
- Percutaneous Transluminal Angioplasty (Active Comparator): The target lesion will be treated by PTA alone.
  Interventions: Device: Percutaneous Transluminal Angioplasty

INTERVENTIONS:
Device: IDEV SUPERA Stent
  Arms: IDEV SUPERA Stent
Device: Percutaneous Transluminal Angioplasty
  Arms: Percutaneous Transluminal Angioplasty

SUMMARY:
Unblinded, randomized, balanced trial comparing 12 month target lesion patency rates of the IDEV SUPERA VERITAS peripheral stent system to PTA in the treatment of obstructive atherosclerotic popliteal artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject has lifestyle limiting claudication or rest pain or at least a single de novo or restenotic popliteal artery lesion.

Exclusion Criteria:

* Intervention distal to the target lesion is required at the time of the index procedure or within 30 days after the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01; Study Completion 2013-01

PRIMARY OUTCOMES:
Primary patency | 12 months
  Primary efficacy will be target lesion primary patency at 12 months.

SECONDARY OUTCOMES:
MAE-free survival rate. | 12 months
  Major Adverse Event-free survival rate that is non-inferior to that of PTA at 12 months.